CLINICAL TRIAL: NCT07163078
Title: A Medical Nutrition Supplement for Cystic Fibrosis
Brief Title: Nutrition Supplement for Cystic Fibrosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Robert DiSilvestro, Emeritus Pofessor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GR134529
Record Dates: First submitted 2025-06-25; First posted 2025-09-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Cystic Fibrosis; Vitamins; Copper; Choline
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional nutrient forms (Active Comparator): People are given a supplement with nutrient forms typically used in supplements
  Interventions: Dietary Supplement: Common form supplementation
- Non-common nutrient forms (Experimental): People are given a supplement with nutrient forms that are not the most commonly used forms in supplements
  Interventions: Dietary Supplement: Uncommon nutrient supplementation

INTERVENTIONS:
Dietary Supplement: Common form supplementation — The intervention product would represent part of a typical supplement given to people including those with CF
  Arms: Conventional nutrient forms
Dietary Supplement: Uncommon nutrient supplementation — The intervention product would represent part of a possible new supplement given to people including those with CF
  Arms: Non-common nutrient forms

SUMMARY:
The goal of this study is to learn if one nutrition supplement formula works better than a different formula in adults with cystic fibrosis. The main question being addressed is: Will certain atypical versions of certain nutrients outperform typical versions of these nutrients? This will be determined by examining blood measures of nutrient levels and/or indications of nutrient function indicators pre- and post-intervention. Participants will take the supplements for 6 weeks with a blood draw before and after that time.

DETAILED DESCRIPTION:
Background. For people with cystic fibrosis (CF), new drugs have extended life expectancy and improved quality of life. Yet, even with these improvements, people with CF still face shorter than normal life spans and constant threats of quality of life disruptions. One approach to attacking these hardships consists of treating nutritional deficiencies. However, that's not as simple as just giving standard nutrients. People with CF have trouble transporting certain nutrients from the digestive system. In theory, giving nutrients in certain forms might get past the CF associated difficulties. However, the big question is: What forms would work?

The answer to this question can vary for different nutrients. For fat soluble vitamins D and E as well as coenzyme Q10 (CoQ10), which is vitamin-like in CF, the proposed solution may be to make the nutrients mix well with water (by using something called micellular versions). That's because these nutrients normally leave the digestive system into the blood by riding with ingested fats; that's a problem in CF because fat malabsorption occurs. Micellular forms could allow the nutrient to travel with water. Some micellular versions of fat soluble vitamins have been tested in people with CF, but the results were not ideal. A better approach could be to use nanoemulsion micellular versions of fat soluble nutrients.

For another nutrient, copper, there needs to not only be good absorption from the digestive system, but also a need to get the copper's to its functional molecules. This principal investigator for the current study has found that giving the normally well absorbed copper glycinate doesn't improve copper status in CF people. In contrast, this situation may be remedied by mixing copper glycinate with a well absorbed version of the nonessential nutrient curcumin (which could escort copper to the appropriate molecules).

Choline, an essential nutrient, can also be a concern for people with CF. Alpha-glyceryl phosphoryl (AGP)-choline may absorb better in these people than the more commonly used choline tartrate.

If the above mentioned non-standard nutrient forms can be shown to work better in people with CF, a new product could be made with the non-standard versions of vitamins D and E, CoQ10, copper, and choline. A formulation could also eventually include another 2 fat soluble vitamins as nanoemulsions as well as zinc + curcumin (since zinc may have the same problem-solution as copper). The product could also include other nutrients normally taken as part of a multi-nutrient supplement.

None of the hand picked versions of the nutrients noted above have been tested in CF people. Therefore, a new study will be done to test these versions for vitamins D and E, CoQ10, copper, and choline.

Hypothesis. This project seeks confirmation of this hypothesis: a formulation with non-standard nutrient versions can outperform conventional nutrients in people with CF. Positive results here can bring a product close to launch. However, one more short study in more people in another geographic location can add more launch justification. A new study can also test the utility of adding 3 nutrients that should work better in versions like those tested in the current project.

Methods. A 6 week intervention is to be used. This principal investigator has used this length in many supplement studies and found it sufficient for altering nutritional function status. For example, this principal investigator has shown a strong change in copper status after 6 weeks of supplementation. Others have seen the same thing for 6 weeks or less for studies on vitamin E.

The new study will be double blind with subjects not knowing whether they are getting the novel or standard nutrient forms. The 2 formulas being tested are as follows:

Supplement 1 Conventional Vitamin D/Vitamin E/Coenzyme Q10. Copper glycinate. Choline tartrate

Supplement 2 Nanoemulsion Vitamin D/ Vitamin E/Coenzyme Q10. Copper glycinate + curcumin. AGP Choline

Daily doses for both supplements 1500 IU Vitamin D3 200; IU Vitamin E; 100 mg Coenzyme Q10; 2.5 mg; 250 mg Choline

Endpoints will be blood assessments for the status of the various nutrients. Some other blood measures will be done that relate to some of the functional implications of improving the status of the nutrients under study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cystic fibrosis
* Diagnosed with exocrine pancreatic insufficiency
* 18 years old or older
* Currently on modulator
* Normal liver enzyme labs

Exclusion Criteria: :

* Non-English-speaking participants
* Acute health crisis
* Persistent elevation of liver enzymes >6 months (E2) (ALT >80 U/L)
* History of liver abnormalities
* If patients are currently taking Category A or Category B in the LiverTox categorization system
* Recent vitamin D supplementation of 30 mcg/day or higher, vitamin E supplements of 200 IU/day or higher, or copper at 2 mg/day or higher
* Any other concern by investigator that the subject is inappropriate for inclusion
* Patients who is on a reduced dose of a CFTR modulator
* Patients on azole antifungals (voriconazole, itraconazole, posaconzole, >7 days of fluconazole, etc.).
* Patients who binge drink EtOH - for men more than 2 drinks/day, for women more than 1 drink/ day
* Patients that are on other medications that are sensitive CYP3A4 substrates - such as tacrolimus for example
* Patients on sensitive CYP3A4 substrates including but not limited to tacrolimus, sirolimus, and cyclosporine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Nutrient status assessor 1 | From pre-supplementation to 6 weeks later
  Plasma concentrations of 25-OH vitamin D (ng/ml)
Nutrition status assessor 2 | From pre-supplementation to 6 weeks later
  Plasma concentrations of vitamin E (mg/L)
Nutrition status assessor 3 | From pre-supplementation to 6 weeks later
  Plasma concentrations of CoQ10 (mg/L)
Nutrition status assessor 4 | From pre-supplementation to 6 weeks later
  Plasma copper (µg/ml)
Nutrition status assessor 5 | From pre-supplementation to 6 weeks later
  Plasma diamine oxidase activity (Units/L)
Nutrition status assessor 6 | From pre-supplementation to 6 weeks later
  Erythrocyte copper superoxide dismutase activities (Units/ml packed cells)
Nutrition status assessor 7 | From pre-supplementation to 6 weeks later
  Plasma choline (µM)

SECONDARY OUTCOMES:
Functional implication indicator 1 | From pre-supplementation to 6 weeks later
  Plasma glucose(mg/dL)
Functional implication indicator 2 | From pre-supplementation to 6 weeks later
  Plasma oxidized LDL (ng/ml)
Functional implication indicator 3 | From pre-supplementation to 6 weeks later
  Plasma alanine amino transferase (ALT)(Units/L)
Functional implication indicator 4 | From pre-supplementation to 6 weeks later
  Plasma vitamin C-like reducing power (mg ascorbic acid equivalents/dL)
Subjective response | From pre-supplementation to 6 weeks later
  Cystic Fibrosis Questionnaire-Revised (CFQ-R): 0-100 scale with higher scores indicating better quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Emeritus Professor, Principal Investigator — Ohio State University; Karen Faculty Pulmonary Medicine Nationwide Children's Hospital, Study Director — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: No
Confidentiality issues exist even if shared without identifiers

REFERENCES:
- [Result] Best K, McCoy K, Gemma S, Disilvestro RA. Copper enzyme activities in cystic fibrosis before and after copper supplementation plus or minus zinc. Metabolism. 2004 Jan;53(1):37-41. doi: 10.1016/j.metabol.2003.07.017. PMID 14681839

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT07163078/Prot_SAP_000.pdf